CLINICAL TRIAL: NCT04682769
Title: Fatigue, Anhedonia and Cardiac Prognostic Markers in Depressed Patients With Coronary Heart Disease
Brief Title: Cardiac Markers in Depressed Patients With Coronary Heart Disease - R01HL147862
Acronym: TREND-3
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: R01HL147862 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Coronary Heart Disease; Depression
MeSH Terms: conditions — Coronary Disease; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with medically stable coronary heart disease and Depressive Disorder
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — Patients with Coronary Heart Disease and Depressive Disorder are receiving routine treatment by their physician.

SUMMARY:
Depression doubles the risk of death in patients with coronary heart disease (CHD), but so far, there is insufficient evidence that we can reduce the risk of death by treating depression. This study will investigate the cardiac risk markers that are associated with depression symptoms that remain despite treatment, and identify potential targets for their treatment. The results of the study will inform the development of more effective interventions to improve both depression and survival in patients with CHD.

DETAILED DESCRIPTION:
Depression is associated with an increased risk of cardiac morbidity and mortality in coronary heart disease (CHD). Although safe and modestly effective treatments for major depression exist, only about 30% of patients ever achieve full remission. CHD patients with depression symptoms that do not respond to treatment are at high risk for cardiac morbidity and mortality compared to those whose depression symptoms respond to treatment. Anhedonia and fatigue are among the most common symptoms to remain following treatment in both depressed CHD patients and in medically well psychiatric patients. In a recent study, the investigators found that several risk markers of cardiovascular morbidity and mortality including a high normal level of the thyroid hormone free thyroxine (FT4), low nocturnal heart rate variability, blunted circadian heart rate, and poor sleep quality predict depression treatment response and post-treatment symptoms of fatigue and anhedonia. It is unclear why these risk markers are associated with residual anhedonia and fatigue. Elevated cortisol levels, chronic sympathetic nervous system activation, reduced vagal modulation of HR, high levels of perceived stress, low level of physical activity, disordered sleep, and occult subclinical thyroid diseases are among the most plausible explanations. Any or all of these factors may explain the relationship between the risk markers and residual fatigue and anhedonia, and all are potentially modifiable and thus possible targets for future clinical trials. The purpose of the proposed research is to identify modifiable correlates of these risk markers and of fatigue and anhedonia in depressed patients with CHD. Study participants will be recruited from cardiology practices at Washington University School of Medicine. Potentially eligible patients will be scheduled for a structured clinical interview. Those who score ≥ 14 on the BDI-II and meet the DSM-5 criteria for major depression and no exclusion criteria will be enrolled. Participants will be evaluated by phone, or in person at the Behavioral Medicine Center at Washington University School of Medicine. The evaluation will be performed in the morning. An appointment will be made for a blood draw on a morning after a 12-hour fast to obtain a thyroid panel, lipid profile, plasma cortisol, C-reactive protein, and other biomarkers. Participants will be fitted with an ambulatory ECG monitor and a wrist actigraph that will be sent to them, and they will complete a battery of self-report inventories. The ECG monitor and actigraph will be worn for 48 hours on two consecutive weekdays to measure the ECG markers, activity levels, and sleep parameters. Participants will be compensated for their time upon return of the samples and equipment. This study will identify potential targets for adjunctive interventions to augment traditional depression treatments and thereby help to lay the groundwork for a randomized clinical trial to determine whether treating depression in patients with CHD can improve both depression and event-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at the Washington University Medical Center with coronary heart disease (CHD) documented by coronary angiography or history of acute coronary syndrome (ACS).
* On a stable medication regimen (only minor changes in drug or dosage in last 30 days) are eligible for recruitment.
* Meet the diagnostic criteria for a depressive disorder, score ≥ 14 on the Beck Depression Inventory (BDI-II), and not meet any exclusion criteria.

Exclusion Criteria:

* Thyroid disease or thyroid medications.
* Moderate to severe cognitive impairment.
* Major psychiatric comorbidities.
* Taking antidepressants other than a selective serotonin reuptake inhibitor (SSRI).
* Suicidal features.
* Current substance abuse.
* New York Heart Association (NYHA) class III or higher or a recent (<3 months) acute coronary syndrome (ACS), coronary artery bypass graft surgery, cardiac hospitalization, or cardiac-related emergency department visit.
* Advanced malignancy, a disability that would prevent compliance with the study protocol, or physician or patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Coronary Disease and Depressive Disorder
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
This is our primary measure of depression severity. | baseline contact
  Beck Depression Inventory (BDI-II)
  scale 0-63; higher score indicates a more severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Freedland, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be shared on request after the closure of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The dataset is expected to be finalized in mid- to late-2025.
Access Criteria: Affiliation with a recognized research institution